CLINICAL TRIAL: NCT01738334
Title: EVALUATION OF THE EFFECTS OF THE MINDFULNESS MEDITATION PRACTICES ON COGNITION OF ADULTS WITH ATTENTION DEFICIT HYPERACTIVITY DISORDER
Brief Title: Effects Of The Mindfulness Meditation Practices On Cognition
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Viviane Freire Bueno, Principal Investigator (Sabine Pompéia), Federal University of São Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMC 001
Record Dates: First submitted 2012-11-11; First posted 2012-11-30 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-11

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Meditation; Cognition; Attention Deficit Disorder with Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Meditation; Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Healthy subjects (Active Comparator): The "active" control group of healthy individuals was subjected to the practice of meditation for eight weeks.
  Interventions: Behavioral: Active comparator (meditation) with healthy subjects
- Standby (No Intervention): The control group of participants (patients and healthy subjects) who was not practice anything for eight weeks.
- Meditation (Experimental): A Group of Patients with ADHD was participate of the meditation practices for eight weeks.
  Interventions: Behavioral: Meditation

INTERVENTIONS:
Behavioral: Active comparator (meditation) with healthy subjects — The control group with healthy subjects that was participate in meditation ("active" control group)
  Arms: Healthy subjects
Behavioral: Meditation — In the eight weeks following the first session of cognitive tests, the participants made a practice of weekly meditation group lasting 2 hours. Practices with each group (patients and "active" controls) occurred on different days. With regard to meditation practices were performed in a sitting posture with emphasis on daily life. Each weekly session involved meditation practices with trained professional, practical proposals for home exercise and a discussion group. Meditation compact discs (CDs)were given to participants for practices at home, which proposed activities for 5 minutes to 1 week and 2 weeks for 10 minutes 3-5, and finally 15 minutes for 6-8 weeks. After 8 weeks of treatment the second session of tests was held that involved the same tasks in session 1.
  Other Names: Mindfulness
  Arms: Meditation

SUMMARY:
Adults with Attention Deficit Hyperactivity Disorder (ADHD) have impairments in attentional subsystems of alerting and conflict monitoring. Mindfulness meditation may lead to an improvement of these deficits, and reduces symptoms of anxiety and depression. However, the studies that demonstrated these improvements did not use a control group, nor controlled the use of medication. In the present study the investigators will examine the effects of the mindfulness practices (same protocol of 8 weekly sessions used in the study that showed positive effects in this disorder) in the performance of adult patients and healthy people (with ADHD). Cognitive performance, mood, and the quality of life will be assessed by validated questionnaires before and after treatment/standby.

ELIGIBILITY:
Inclusion Criteria:

* Portuguese as their first language;
* minimum of eight years of formal education;
* normal vision or corrected to normal and normal hearing;
* no prior experience with meditation;
* patients should be taking stable doses of methylphenidate (for at least a month) for their disorder as prescribed by their doctors.

Exclusion Criteria:

* patients with neurological and psychiatric disorders such as psychosis, obsessive-compulsive disorder or Tourette's syndrome.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-02; Primary Completion 2012-02 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Evaluate the ADHD symptoms before to the meditation and after 8 weeks to the meditation. | change from baseline in ADHD symptoms at 8 weeks
  The symptoms of inattention and hyperactivity / impulsivity were evaluated by means the Adult self-report scale (ASRS).
Evaluate the executive functions | 1 day
  The executive functions tests were applied before to the meditation, so that to avoid learning.
Evaluate the mood symptoms before to the meditation and 8 weeks after to the meditation. | change from baseline in mood symptoms at 8 weeks.
  The symptoms of anxiety and depression were evaluated by means of the following scales: Trait Anxiety Inventory (STAI-Trait), and Beck Depression Scale, respectively, and the visual-analog scales of mood (VAMS)and Positive and negative Affect Schedule extended (PANAS-X).
Evaluate the quality of life before to the meditation and 8 weeks after to the meditation. | change from baseline in quality of life at 8 weeks.
  Quality of Life was evaluated by means of the Questionnaire in Adults with ADHD (AAQoL).
Evaluate the attention before to the meditation and 8 weeks after to the meditation. | change from baseline in attention at 8 weeks.
  The scores of attention was evaluated by Continuous Performance Test (CPT) and the Attentional Network Test (ANT).

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Pompéia, Postdoctoral, Study Director — Federal University of São Paulo; Viviane F Bueno, Doctor, Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of São Paulo, São Paulo, São Paulo, Brazil